CLINICAL TRIAL: NCT01906372
Title: Open Label Proof of Concept Study to Evaluate Efficacy and Safety of Adrenocorticotropic Hormone Gel in Refractory Dermatomyositis or Polymyositis
Brief Title: Acthar in Treatment of Refractory Dermatomyositis and Polymyositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rohit Aggarwal, MD (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Rohit Aggarwal, MD, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO13050507
Record Dates: First submitted 2013-07-05; First posted 2013-07-24 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Dermatomyositis; Polymyositis
Keywords: dermatomyositis; polymyositis
MeSH Terms: conditions — Dermatomyositis; Polymyositis

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acthar Gel (Experimental): Acthar Gel (Adrenocorticotropic Hormone Gel)in refractory PM and DM patients using an open label design for 6 months. We will enroll 10 active and refractory PM/DM patients over a 15 month period, followed by 6 months of additional follow-up for each subject. Study subjects will self-administer subcutaneously H.P. Acthar Gel 80 units (1 ml) twice a week for a period of six months. Outcome measures were not evaluated on subjects who did not reach the 8 week time point in the trial.
  Interventions: Drug: Adrenocorticotropic Hormone Gel

INTERVENTIONS:
Drug: Adrenocorticotropic Hormone Gel — H.P. Acthar Gel 80 units will be self-administered subcutaneously twice weekly by the subject for a period of 6 months.
  Other Names: H.P. Acthar Gel

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of the study drug, ACTH Gel in people diagnosed with dermatomyositis a disease that causes muscle weakness and is associated with a rash (DM) or polymyositis (PM) a disease that causes muscle weakness without a rash. The study doctors want to evaluate whether ACTH Gel will improve the symptoms of this disease. This drug is approved by the Food and Drug Administration (FDA) for dermatomyositis (DM) and polymyositis (PM). ACTH gel has been an FDA-approved treatment for myositis since 1952, and in 2010 the FDA retained PM and DM as diseases approved for ACTH gel use.

DETAILED DESCRIPTION:
Despite its FDA approval there is very limited data on its clinical effectiveness in PM and DM. There was a recent study published in the peer-review journal Drug Design, Development and Therapy on a retrospective case series evaluating Acthar in the treatment of PM and DM. Acthar was administered to five patients who had previously failed multiple steroid and immunosuppressant treatment regimens. The patients received injections of Acthar over the course of 12 weeks or more. Improvement in PM and DM symptoms related to disease exacerbations was seen in all five patients. Symptom improvements included increased muscle strength, resolution of disease-related skin manifestations and improvements in the ability to perform tasks associated with daily living. All of these patients tolerated the treatment well with no significant side effects reported. The paper, "Treating refractory dermatomyositis or polymyositis with adrenocorticotropic hormone gel: a retrospective case series," was authored by Dr. Todd Levine, M.D., Co-Director of the Neurophysiology Department at Banner Good Samaritan Medical Center, Assistant Professor at the University of Arizona in Neurology, and Member of Phoenix Neurological Associates.

H.P. Acthar® Gel, or Acthar, is a prescription medication containing the hormone adrenocorticotropin (hormone produced and secreted by the anterior pituitary gland), also known as ACTH. H.P. Acthar Gel is a highly purified preparation of adrenocorticotropic hormone (ACTH) in a gel that is designed to provide extended release of the ACTH following injection. Acthar was originally approved by the FDA in 1952. It is approved for use in 19 different conditions including dermatomyositis and polymyositis.

Acthar is designed to provide a prolonged release of the medication after it is injected. Acthar is not a steroid; it works by helping your body produce its own natural steroid hormones, such as cortisol, corticosterone, and aldosterone. Acthar is an injection that is given intramuscularly (into the muscle). Subjects enrolled in the study will be asked to self administer Acthar two times per week. Subjects will be provided training by the principal investigator on how to perform the self injections.

ELIGIBILITY:
Inclusion Criteria:

* Definite or probable polymyositis (PM) or dermatomyositis (DM) by Bohan and Peter criteria.
* PM patients must either possess a myositis-associated autoantibody or undergo adjudication for confirmation of the PM diagnosis by consensus of two experts to ensure non-PM patients are not enrolled. This step is necessary since there are well-known mimics of PM.
* Age ≥ 18 years.
* Active myositis as defined by baseline Manual Muscle Testing (MMT-8) no greater than 125/150 and at least 2 additional CSM meeting the criteria stipulated below:

  1. Patient global with a minimum value of 2.0 cm on a 10 cm visual analog scale(VAS)
  2. Physician global with a minimum value of 2.0 cm on a 10 cm VAS scale
  3. Health Assessment Questionnaire (HAQ) disability index with a minimum value of 0.25
  4. Elevation of at least one of the muscle enzymes [which includes creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] at a minimum level of 1.3 x the upper limit of normal.
  5. Global extramuscular disease activity score with a minimum value of 1.0 cm on a 10 cm VAS scale [this measure is the physician's composite evaluation and is based on assessments of activity scores on the constitutional, cutaneous, skeletal, gastrointestinal, pulmonary and cardiac scales of the Myositis Disease Activity Assessment Tool (MDAAT)].
* To ensure that we can enroll active DM patients with a severe rash who may not meet the MMT-8 criterion noted above, we propose additional enrollment criteria such that the International Myositis Assessment and Clinical Studies (IMACS) definition of improvement (DOI) can potentially be met:

  1. Cutaneous VAS score on MDAAT > 3 cm on a 10 cm VAS scale, and
  2. At least 3 of the above 5 (a through e under 4.) criteria.
* Refractory myositis is defined by active disease despite an adequate glucocorticoid trial (> 2 months of usual glucocorticoid therapy or intolerance to such therapy) and/or ≥ 1 conventional immunosuppressive agent (e.g. methotrexate, azathioprine, tacrolimus, cyclosporine, mycophenolate mofetil, IVIG, anti-TNF or rituximab) for a reasonable dose and duration (> 3 months or intolerance to therapy). It is recommended to enroll refractory patients failing (or intolerant to) both glucocorticoids and at least 1 conventional immunosuppressive agent.
* If the enrolling physician is planning to continue current immunosuppressive agents or glucocorticoids as concomitant therapy with Acthar gel during the trial, then patient must be on a stable glucocorticoid and/or immunosuppressive dose 2 weeks prior to visit 1. The patient should have been on that immunosuppressive medication for at least 8 weeks (and at least 4 weeks for glucocorticoids) prior to visit 1.
* If the enrolling physician is planning to discontinue current immunosuppressive agent or glucocorticoids, then following wash out period is required prior to visit 1.
* If previous concomitant medications were discontinued, the following wash out periods are required prior to Visit 1
* Methotrexate -4 weeks
* Other IS agent (e.g. azathioprine, cyclosporine, tacrolimus, leflunomide, mycophenolate mofetil) - 4 weeks
* IVIg or cyclophosphamide - 2 months
* rituximab -6 months
* infliximab or adalimumab -8 weeks
* glucocorticoids - 2 weeks
* etanercept -2 weeks
* anakinra -1 week

Exclusion Criteria:

* Juvenile DM or PM, myositis in overlap with another connective tissue disease, cancer associated myositis, inclusion body myositis, or any other non immune-mediated myopathy.
* Hypersensitivity to Acthar
* Severe cardiac or pulmonary involvement
* Severe muscle damage defined as a baseline global muscle damage score on the MDI (Myositis Damage Index) of ≥ 5 cm on a 10 cm VAS.
* Patients with malignancy within 3 years of screening (except basal cell cancer or squamous cell cancer of skin).
* Uncontrolled diabetes, hepatic or renal disease.
* Ongoing active or chronic infections.
* Pregnant or lactating females.
* For any medical or physical or socio-psychological reasons that PI feels would not allow the subject to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Aggarwal, MD, Principal Investigator — University of Pittsburgh, Division of Rheumatology
Locations (2):
- United States (2):
  - North Shore LIJ Medical Center, Great Neck, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catania A, Gatti S, Colombo G, Lipton JM. Targeting melanocortin receptors as a novel strategy to control inflammation. Pharmacol Rev. 2004 Mar;56(1):1-29. doi: 10.1124/pr.56.1.1. PMID 15001661
- [Background] Catania A, Lonati C, Sordi A, Carlin A, Leonardi P, Gatti S. The melanocortin system in control of inflammation. ScientificWorldJournal. 2010 Sep 14;10:1840-53. doi: 10.1100/tsw.2010.173. PMID 20852827
- [Background] Baram TZ, Mitchell WG, Tournay A, Snead OC, Hanson RA, Horton EJ. High-dose corticotropin (ACTH) versus prednisone for infantile spasms: a prospective, randomized, blinded study. Pediatrics. 1996 Mar;97(3):375-9. PMID 8604274
- [Background] Bomback AS, Tumlin JA, Baranski J, Bourdeau JE, Besarab A, Appel AS, Radhakrishnan J, Appel GB. Treatment of nephrotic syndrome with adrenocorticotropic hormone (ACTH) gel. Drug Des Devel Ther. 2011 Mar 14;5:147-53. doi: 10.2147/DDDT.S17521. PMID 21448451
- [Background] Simsarian JP, Saunders C, Smith DM. Five-day regimen of intramuscular or subcutaneous self-administered adrenocorticotropic hormone gel for acute exacerbations of multiple sclerosis: a prospective, randomized, open-label pilot trial. Drug Des Devel Ther. 2011;5:381-9. doi: 10.2147/DDDT.S19331. Epub 2011 Jul 11. PMID 21792296
- [Background] Levine T. Treating refractory dermatomyositis or polymyositis with adrenocorticotropic hormone gel: a retrospective case series. Drug Des Devel Ther. 2012;6:133-9. doi: 10.2147/DDDT.S33110. Epub 2012 Jun 11. PMID 22787386
- [Background] Rider LG, Giannini EH, Brunner HI, Ruperto N, James-Newton L, Reed AM, Lachenbruch PA, Miller FW; International Myositis Assessment and Clinical Studies Group. International consensus on preliminary definitions of improvement in adult and juvenile myositis. Arthritis Rheum. 2004 Jul;50(7):2281-90. doi: 10.1002/art.20349. PMID 15248228
- [Background] Oddis CV, Reed AM, Aggarwal R, Rider LG, Ascherman DP, Levesque MC, Barohn RJ, Feldman BM, Harris-Love MO, Koontz DC, Fertig N, Kelley SS, Pryber SL, Miller FW, Rockette HE; RIM Study Group. Rituximab in the treatment of refractory adult and juvenile dermatomyositis and adult polymyositis: a randomized, placebo-phase trial. Arthritis Rheum. 2013 Feb;65(2):314-24. doi: 10.1002/art.37754. PMID 23124935
- [Derived] Fernandez AP, Gallop J, Polly S, Khanna U. Efficacy and safety of repository corticotropin injection for refractory cutaneous dermatomyositis: a prospective, open-label study. Rheumatology (Oxford). 2024 Dec 1;63(12):3370-3379. doi: 10.1093/rheumatology/kead595. PMID 37941470
- [Derived] Aggarwal R, Marder G, Koontz DC, Nandkumar P, Qi Z, Oddis CV. Efficacy and safety of adrenocorticotropic hormone gel in refractory dermatomyositis and polymyositis. Ann Rheum Dis. 2018 May;77(5):720-727. doi: 10.1136/annrheumdis-2017-212047. Epub 2017 Dec 13. PMID 29237618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with active and refractory polymyositis or dermatomyositis were recruited at two clinical centers, The University of Pittsburgh and North Shore Long Island Jewish Center over a 16 month recruitment period. Two subjects did not reach the week 8 time point prior to withdrawing from the trial therefore additional subjects were enrolled.
Pre-assignment Details: If the enrolling physician planned to discontinue a specific immunosuppressive agent or glucocorticoid prior to study visit 1, a pre-defined washout period was required.
Groups:
- Acthar Gel: Acthar Gel (Adrenocorticotropic Hormone Gel) 80 units (1 ml) twice a week for a period of six months.
Period: Overall Study
Arm/Group | Acthar Gel
Started | 12
Visit 7: Treatment Phase Completed | 10
Visit 10: Follow up Phase Completed | 8
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: A total of 12 participants were enrolled however only 11 participants were assessed for baseline characteristics due to one subject withdrawing after screening and never received study drug.
Groups:
- Acthar Gel: Acthar Gel (Adrenocorticotropic Hormone Gel)in refractory PM and DM patients using an open label design for 6 months. Study subjects will self-administer subcutaneously H.P. Acthar Gel 80 units (1 ml) twice a week for a period of six months.
Arm/Group | Acthar Gel
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Diagnosis [Count of Participants; unit: Participants]
  Dermatomyositis | 6
  Polymyositis | 5
Disease Duration [Mean (Standard Deviation); unit: years] — Population: One additional patient dropped out of the study at 6 weeks due to worsening of conduction abnormalities (heart block unrelated to the study drug), since the patient had not completed minimum 8 weeks of study drug required for outcome assessment as per study protocol, he was not included in primary analysis.
  years
    number analyzed (Participants) | 10
    (all) | 2.0 (2.0)
Autoantibody Status [Count of Participants; unit: Participants] — Population: One additional patient dropped out of the study at 6 weeks due to worsening of conduction abnormalities (heart block unrelated to the study drug), since the patient had not completed minimum 8 weeks of study drug required for outcome assessment as per study protocol, he was not included in primary analysis.
  Participants
    number analyzed (Participants) | 10
    (all) | 8

OUTCOME MEASURES:

1. Primary Outcome: Specific Aim 1: Number of Subjects Meeting IMACS Preliminary Definition of Improvement (DOI).
Description: 3 of any of the 6 core set measures (CSM) improved by ≥ 20%, with no more than 2 CSM worsening by ≥25% (worsening measure cannot include the MMT). The DOI should be met at least once on any of the 6 follow up visits and maintained until week 24. Subjects not meeting DOI during the trial are treatment failures.
Time Frame: Primary end point: IMACS preliminary definition of improvement (DOI)
Population: Total of 10 PM/DM patients completed the study.One additional patient dropped out of the study at 6 weeks due to worsening of conduction abnormalities (heart block unrelated to the study drug).The patient had not completed minimum 8 weeks of study drug required for outcome assessment as per study protocol, and was not included in primary analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Acthar Gel: Acthar Gel (Adrenocorticotropic Hormone Gel) in active and refractory PM and DM patients using an open label design for 6 months. Study subjects self-administered subcutaneously H.P. Acthar Gel 80 units (1 ml) twice a week subcutaneously for a period of six months.
Arm/Group | Acthar Gel
Number analyzed (Participants) | 10
Participants | 7
Statistical Analysis 1: Comparison: Acthar Gel; Test type: Superiority or Other; Open label single arm pilot trial without control group; Frequency of achieving primary endpoint = 0.70

2. Secondary Outcome: Steroid-sparing Effect of H.P. Acthar Gel in Refractory Adult PM and DM Patients.
Description: Mean change in glucocorticoid dose (equivalent prednisone dose) at 24 weeks compared to baseline.
Time Frame: Steroid sparing effect and safety and tolerability at 24 weeks compared to baseline
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Acthar Gel: Acthar Gel (Adrenocorticotropic Hormone Gel)in refractory PM and DM patients using an open label design for 6 months. 10 active and refractory PM/DM patients were evaluated over a 15 month period, followed by 6 months of additional follow-up for each subject. Study subjects will self-administer subcutaneously H.P. Acthar Gel 80 units (1 ml) twice a week for a period of six months.
Arm/Group | Acthar Gel
Number analyzed (Participants) | 10
mg
  Follow Up 24 weeks | 2.3 (3.2)
  Baseline | 18.5 (15.7)
Statistical Analysis 1: Comparison: Acthar Gel; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the overall duration of the study (12 months).
Description: Adverse events with a causality of possibly, probably or definitely related to medicinal product at included in this reporting data.
Arm/Group | Acthar Gel
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acthar Gel (N=10)
Avascular Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Subject hospitalized for a total left hip arthroplasty which confirmed diagnosis of avascular necrosis. Site investigator reported this event as probably related to study drug.
Local infection with moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, a (Infections and infestations) | 2 (2) — One subject with diagnosis of disseminating herpes zoster and one subject with herpes zoster infection. Both subjects received IV antivirals.
Atrioventricular Block (Cardiac disorders) | 1 (1) — Subject was hospitalized for a third degree AV heart block with subsequent transvenous pacemaker placed. The site investigator reported this event as not related to study drug.
Non-cardiac chest pain (General disorders) | 1 (1) — Subsequent testing ruled out cardiac event. Discharge diagnosis of chest pain most likely musculoskeletal. Site investigator reported this event as unlikely related to study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acthar Gel (N=10)
Sinus Tachycardia (Cardiac disorders) | 1 (1) — Sinus tachycardia confirmed by electrocardigram. PI feels that this is likely related to the SAE of dissemenated herpes zoster infection which was deemed possibly related to study drug.
Diarrhea (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions (General disorders) | 4 (4) — Bruising at injection site.
Sinusitis (Infections and infestations) | 1 (1)
Upper Respiratory Infections (Infections and infestations) | 1 (1)
Cholesterol high (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) — Subject reported worsening of anxiety symptoms.
Agitation (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Lung nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Chest x-ray and computerized tomography scan revealed nodules in both lungs. Chest x-ray from 5 days earlier was unremarkable. Lung biopsy was done and tests confirmed the pulmonary nodules were most likely caused by the herpes zoster virus.
Calcinosis (Skin and subcutaneous tissue disorders) | 2 (2) — One subject with subtle worsening of the subcutaneous calcinosis confirmed on imaging studies. One subject with significant new calcification in left breast which were not present prior to Acthar administration.
Hypertension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Small pilot open label single arm trial. Larger double blinded placebo controlled randomized trials are required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No